CLINICAL TRIAL: NCT01773096
Title: The Use of Methylnaltrexone to Reduce Post-operative Opioid-induced Constipation in the Pediatric Spinal Fusion Patient
Brief Title: Methylnaltrexone Use for Opioid-induced Postoperative Constipation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shriners Hospitals for Children (Other)
Responsible Party: Principal Investigator, Deborah J. Vermaire MD, Anesthesiologist, Shriners Hospitals for Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MNTX-2013
Record Dates: First submitted 2013-01-15; First posted 2013-01-23 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Constipation
Keywords: opioid-induced
MeSH Terms: conditions — Constipation | interventions — methylnaltrexone; Sennosides; Dioctyl Sulfosuccinic Acid; Bisacodyl; Magnesium Hydroxide; polyethylene glycol 3350; Polyethylene Glycols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study group (Experimental): Weight-based dose (0.15 mg/kg for patients less than 38 kg, 8 mg for patients weighing 38-62 kg, or 12 mg for patients weighing greater than 62 kg) of methylnaltrexone will be administered on post-operative day 3 and again, if indicated, on post-operative day 4. This group will also receive the standard bowel protocol beginning on postoperative day one as per protocol.
  Interventions: Drug: Methylnaltrexone; Drug: Senna, docusate sodium, bisacodyl, magnesium hydroxide, Miralax
- Institutional bowel protocol (Active Comparator): Patient will receive institutional standard bowel protocol. Beginning on post-operative day one either miralx,docusate sodium or senna, on a weight-based dose. If no bowel movement in 72 hours, either oral bisacodyl or magnesium hydroxide, on a weight-based dosing, will be added.
  Interventions: Drug: Senna, docusate sodium, bisacodyl, magnesium hydroxide, Miralax

INTERVENTIONS:
Drug: Methylnaltrexone — Patient will receive methylnaltrexone on postoperative day 3 on a weight based dose and again 24 hours later if required.
  Other Names: Relistor
  Arms: Study group
Drug: Senna, docusate sodium, bisacodyl, magnesium hydroxide, Miralax — Standard institutional bowel protocol will begin on post-operative day 1. Miralax,Docusate sodium or senna will be given on a weight-based dosing. If no bowel movement in 72 hours, bisacodyl or magnesium hydroxide will be added.
  Other Names: Senokot,Colace, Dulcolax, Milk of Magnesia, polyethylene glycol

SUMMARY:
The purpose of this study is to determine whether the routine use of methylnaltrexone in the post-operative pediatric spinal fusion patient will decrease the incidence of constipation.

DETAILED DESCRIPTION:
Methylnaltrexone will be given to pediatric patients post-operative from spinal fusion surgery on post-operative day number 3 and then again on postoperative day number 4, if no laxation achieved. Various outcome measures, safety and efficacy of the drug will be observed and recorded.

ELIGIBILITY:
Inclusion Criteria:

* spinal fusion surgery
* current opioid use
* 12 years of age and older
* no or inadequate bowel movement by post-operative day 3

Exclusion Criteria:

* known or expected mechanical bowel obstruction
* known or suspected lesions of the GI tract
* unexpected transfer to ICU
* unexpected return to the operating room
* patient or parent refusal of methylnaltrexone
* incomplete data concerning time to laxation

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
reduction of post-operative opioid induced constipation | first post-operative week

SECONDARY OUTCOMES:
time to ambulation in post-operative pediatric spinal fusion patients | first post-operative week

OTHER OUTCOMES:
time to oral intake of pediatric post-operative spinal fusion patient | first post-operative week

CONTACTS AND LOCATIONS:
Overall Officials: Deborah J. Vermaire, M.D., Principal Investigator — Shriners Hospitals for Children
Locations (1):
- Shriners Hospitals for Children- Spokane, Spokane, Washington, United States

REFERENCES:
- [Result] Anissian L, Schwartz HW, Vincent K, Vincent HK, Carpenito J, Stambler N, Ramakrishna T. Subcutaneous methylnaltrexone for treatment of acute opioid-induced constipation: phase 2 study in rehabilitation after orthopedic surgery. J Hosp Med. 2012 Feb;7(2):67-72. doi: 10.1002/jhm.943. Epub 2011 Oct 13. PMID 21998076